CLINICAL TRIAL: NCT07106463
Title: Microbiota: Its Role in Chronic Inflammation, IDB and Risk of Colorectal Cancer. Evaluation of a Predictive Prognostic Model With Therapeutic Implications
Status: Active, not recruiting | Type: Observational
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Massimiliano Berretta, Full Professor of Medical Oncology, University of Messina
Other Study IDs: 07-24
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: IBD (Inflammatory Bowel Disease); Colon Cancer
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months

SUMMARY:
The gut microbiome is emerging as a crucial factor in several intestinal diseases, contributing to the etiopathogenesis of inflammatory disorders. While most microorganisms reside in the gut and play vital roles in host immunity and nutrition, an imbalance in microbiome composition can trigger chronic intestinal inflammation, increasing the risk of developing colorectal cancer (CRC). Significant quantities of the Gram-negative bacterium Fusobacterium nucleatum have been associated with poorer survival rates and increased resistance to chemotherapy in CRC patients. Furthermore, F. nucleatum has been shown to mediate CRC chemoresistance through activation of the ULK1 autophagy pathway. Recent studies have reported the ability of F. nucleatum to induce inflammation in the gut epithelium and activate a specific component of the immune system, the NLRP3 inflammasome, leading to the release of IL-1ß, a pro-inflammatory cytokine. The aim of this project is to investigate the role of F. nucleatum in the development of chronic inflammatory bowel disease (IBD) and CRC by exploring a potential connection between its involvement in NLRP3 inflammasome activation and its ability to promote chemoresistance through autophagy modulation. The working hypothesis posits that these two biological processes are strongly interconnected and may significantly influence the interaction between the gut microbiota and host immunity, ultimately affecting disease progression in IBD and CRC. The proposed research plan includes:

i) in vitro characterization of the impact of F. nucleatum infection on NLRP3 inflammasome activation, autophagy induction, and CRC development and progression; ii) determination of the correlation between F. nucleatum abundance and chronic IBD, as well as early and advanced stages of colorectal carcinomas; iii) implementation of radiomic analyses to accurately distinguish cancerous from non-cancerous colon tissue and to identify radiomic signatures indicative of specific tumor-host interactions, including inflammation and/or autophagy. This research aims to generate novel insights into the interplay between the microbiota and chronic degenerative diseases, thereby contributing to the development of innovative microbiota-based therapeutic strategies. This proposal may represent an effective approach to predict patient outcomes and improve the prognosis of individuals with IBD and CRC by enabling differential patient management, correlating F. nucleatum levels with inflammation and autophagy, and potentially informing combinatorial treatments to overcome chemoresistance.

ELIGIBILITY:
Inclusion Criteria:

Individuals in generally good health

Individuals diagnosed with Inflammatory Bowel Disease (IBD)

Individuals diagnosed with early-stage Colorectal Cancer (CRC)

Individuals with locally advanced Colorectal Cancer (CRC)

Individuals with metastatic Colorectal Cancer (CRC)

Exclusion Criteria:

Individuals diagnosed with other malignancies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: individuals in health, with IBD, with early CRC, with local advanced CRC and metastatic CRC (20 subjects for arms).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
Levels of NLRP3 inflammasome activation, autophagy markers, and colorectal cancer-related molecular changes in in vitro models infected with F. nucleatum. | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Quantification of F. nucleatum levels in biological samples from individuals with chronic inflammatory bowel disease and colorectal carcinomas. | Baseline

OTHER OUTCOMES:
Correlation between CT-derived radiomic features, histological findings, F. nucleatum abundance, and inflammation markers in patients with varying levels of intestinal inflammation. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria "G.Martino", Messina, Italy, Italy